CLINICAL TRIAL: NCT05721898
Title: Assessment of Cortical Bone Mechanics Technology (CBMT) Fracture Discrimination Capability
Acronym: STRONGER
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Collaborators: Indiana University School of Medicine (Other); University of Florida (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Brian Clark, Professor, Ohio University
Other Study IDs: 21-F-1
Record Dates: First submitted 2023-01-28; First posted 2023-02-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis; Osteopenia or Osteoporosis; Osteoporosis, Postmenopausal; Osteoporosis Risk; Osteoporotic Fractures; Fragility Fracture; Bone Fracture
Keywords: Osteoporosis; Bone strength; Fracture
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Osteoporotic Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fracture Cases: Fragility Fracture Cases: Post-menopausal females between 50-80 years who have experienced a fragility fracture of the arms (including wrist fractures) or legs (including hip, pelvis, or ankle fractures) after the age of 50 years. Fractures of the spine, digits, toes or face will not be considered. A fragility fracture is operationally define based on self-report of an arm or leg fracture caused by falls from a height <6 inches. A fragility fracture will not count if it is associated with 1) running, bicycling or other similar fast-moving activity such as sports subjects, 2) being struck by a falling or otherwise quickly moving heavy object, or 3) a motor vehicle accident. Insufficiency/stress fractures will not be included. Body mass index between 18.5 and 35 kg/m2.
  Interventions: Diagnostic Test: Cortical Bone Mechanics Technology
- Non-Fracture Controls: Controls: Post-menopausal females between 50-80 years who have not experienced a fracture at any site after the age of 40 years (does not include fractures of the digits, toes or face). Does not self-report losing more than 1.5 inches in stature (height) in the previous 15 years. Body mass index between 18.5 and 35 kg/m2.
  Interventions: Diagnostic Test: Cortical Bone Mechanics Technology

INTERVENTIONS:
Diagnostic Test: Cortical Bone Mechanics Technology — Cortical Bone Mechanics Technology (CBMT). CBMT testing will be performed bilaterally, and flexural rigidity (EI) will be calculated. If a participant has fractured a wrist or forearm bone in the prior 1-year, then only the arm that was not fractured will be tested. During testing, participants will lie supine in the CBMT instrument.

SUMMARY:
Osteoporosis is a disease characterized by low bone mass and structural deterioration of bone tissue leading to bone fragility (i.e., weakness) and an increased risk for fracture. Bone strength is a critical factor in a bone's ability to resist fracture and is clearly an important outcome in studies of osteoporosis. The current standard for assessing bone health and diagnosing osteoporosis is to use dual-energy x-ray absorptiometry (DXA) to quantify the areal bone mineral density (BMD), typically at the hip and spine. However, DXA-derived BMD has limited discriminatory accuracy for distinguishing individuals that experience fragility fracture from those who do not. One well known limitation of DXA-derived BMD is that it does not adequately assay bone strength. There is a critical unmet need to identify persons more accurately with diminished bone strength who are at high risk of experiencing a fragility fracture in order to determine an appropriate therapy. A potential new diagnostic approach to assess skeletal health and improve osteoporosis diagnosis is the use of Cortical Bone Mechanics Technology (CBMT). CBMT leverages multifrequency vibration analysis to conduct a noninvasive, dynamic 3-point bending test that makes direct, mechanical measurements of ulnar cortical bone. Data indicates that CBMT-derived ulnar flexural rigidity accurately estimates ulnar whole bone strength and provides information about cortical bone that is unique and independent of DXA-derived BMD. However, the clinical utility of CBMT-derived flexural rigidity has not yet been demonstrated. The investigators have designed a clinical study to assess the accuracy of CBMT-derived ulnar flexural rigidity in discriminating post-menopausal women who have suffered a fragility fracture from those who have not. These data will be compared to DXA-derived peripheral and central measures of BMD obtained from the same subjects.

DETAILED DESCRIPTION:
Osteoporosis is a disease characterized by low bone mass and structural deterioration of bone tissue, leading to bone fragility (i.e., weakness), and an increased risk for fracture. The incidence of osteoporosis related fragility fractures (i.e., low energy fractures resulting from a fall from standing height or less) increases with age and is highest in post-menopausal women. In the United States, there were approximately 2.3 million fragility fractures in 2020. The total annual expense of providing direct and indirect care for osteoporotic fractures among Medicare beneficiaries was estimated at $57 billion in 2018, with an expected increase to over $95 billion by 2040.

Bone strength is a critical factor in a bone's ability to resist fracture and is clearly an important outcome in studies of osteoporosis. The current standard for assessing bone health and diagnosing osteoporosis is to use dual-energy x-ray absorptiometry (DXA) to quantify the areal bone mineral density (BMD), typically at the hip and spine. However, DXA-derived BMD has relatively poor discriminatory accuracy to distinguish individuals who will fracture from those who will not.

One well known limitation of BMD is that it does not adequately assay bone strength. As with any complex structure, bone strength depends on the interplay between a variety of factors, including the amount or mass of bone present and the structural organization and quality of the material. BMD primarily indicates bone mass but does not adequately assess the contributions of bone structure or quality to bone strength.

Reflecting the limitations of DXA, BMD explains less than half of the variation in whole bone strength, and when bone strength is improved and fracture risk reduced via bisphosphonate drug therapy, less than 18% of the observed reductions in vertebral fracture risk can be attributed to increases in BMD. These findings clearly suggest that the current standard care is insufficient for identifying those who might benefit most from early intervention to improve bone health, as well as for assessing the effect of new therapies targeted at increasing bone strength. A potential new diagnostic approach to address this critical unmet need and improve osteoporosis diagnosis is the use of Cortical Bone Mechanics Technology (CBMT).

CBMT leverages multifrequency vibration analysis to conduct a noninvasive, dynamic 3-point bending test that makes direct, functional mechanical measurements of ulnar cortical bone (e.g., flexural rigidity). Because CBMT is a whole bone test, its measurements reflect the combined influences of bone quantity, structure, and quality at all hierarchical levels. Its validity in accurate measurements of ulna flexural rigidity and estimations of quasistatic ulna bending strength have been demonstrated. CBMT-derived flexural rigidity yielded a near perfect estimate of cadaveric bone strength (R2=0.99). Additionally, flexural rigidity has been reported to decrease 21% following potassium hydroxide-induced collagen degradation whereas BMD was not altered. Thus, current data indicates that CBMT-derived ulnar flexural rigidity accurately estimates ulnar whole bone strength and provides information about cortical bone that is unique and independent of BMD. Assessing cortical bone, in particular, is important because after ~65 years most bone loss is cortical, and the cortical bone loss is associated with increased incidence of fragility fractures. However, the clinical utility of CBMT-derived flexural rigidity has not yet been demonstrated.

The investigators have designed a clinical study to assess the accuracy of CBMT-derived ulnar flexural rigidity in discriminating post-menopausal women who have suffered a fragility fracture from those who have not. These data will be compared to DXA-derived peripheral and central measures of BMD obtained from the same subjects.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Subjects Who Have Experienced a Fragility Fracture (Cases) Inclusion Criteria

* Female.
* Age range: 50 to 80 years at recruitment. All subjects must self-report that their last menses occurred at least 24-months prior to enrollment.
* Has experienced a fragility fracture of the arms (including wrist fractures) or legs (including hip, pelvis, or ankle fractures) after the age of 50 years. Fractures of the spine, digits, toes or face will not be considered. A fragility fracture is operationally define based on self-report of an arm or leg fracture caused by falls from a height <6 inches. A fragility fracture will not count if it is associated with 1) running, bicycling or other similar fast-moving activity such as sports subjects, 2) being struck by a falling or otherwise quickly moving heavy object, or 3) a motor vehicle accident. Insufficiency/stress fractures will not be included.
* Body mass index between 18.5 and 35 kg/m2.
* Physically able to safely participate in the study activities.
* Able to provide informed consent.

Exclusion Criteria

* Failure to provide informed consent.
* Has had bilateral hip replacements.
* Lives in a nursing home; persons living in assisted or independent housing will not be excluded.
* Self-reported type 1 diabetes.
* Unable to communicate because of severe hearing loss or speech disorder.
* Self-reports being told by a physician that they have a terminal illness.
* The subject will be excluded if they answer yes to the following question: Do you have an active rotator cuff tear, had shoulder surgery in the past 12-months, or experience severe shoulder, wrist, or elbow joint pain on a regular basis?
* Use of systemic glucocorticoids for more than 6-months in the prior one year.
* Self-reported diseases that could interfere with bone metabolism. For example, osteomalacia, bone cancer, myeloma, Pagets disease, hyper parathyroidism, hyperthyroidism not treated, severe renal (stage 4+ chronic kidney disease, history of dialysis, kidney transplant, etc.) or hepatic insufficiency, prolonged immobilization (more than 2 months in the previous year).
* If, in the opinion of a site PI, the subject is inappropriate for the scientific purposes of this study. For instance, a high fall risk patient due to an existing neurological disorder (e.g., Parkinsons disease, ALS, etc.) would be excluded.

Inclusion and Exclusion Criteria for Subjects Who Have Not Experienced a Fragility Fracture (Controls) Inclusion Criteria

* Female.
* Age range: 50 to 80 years at recruitment. All subjects must self-report that their last menses occurred at least 24-months prior to enrollment.
* Self-reports not experiencing a fracture at any site after the age of 40 years (does not include fractures of the digits, toes or face).
* Does not self-report losing more than 1.5 inches in stature (height) in the previous 15 years.
* Body mass index between 18.5 and 35 kg/m2.
* Physically able to safely participate in the study activities.
* Able to provide informed consent.

Exclusion Criteria

* Failure to provide informed consent.
* Has had bilateral hip replacements.
* Lives in a nursing home; persons living in assisted or independent housing will not be excluded.
* Self-reported type 1 diabetes.
* Unable to communicate because of severe hearing loss or speech disorder.
* Self-reports being told by a physician that they have a terminal illness.
* The subject will be excluded if they answer yes to the following question: Do you have an active rotator cuff tear, had shoulder surgery in the past 12-months, or experience severe shoulder, wrist, or elbow joint pain on a regular basis?
* Use of systemic glucocorticoids for more than 6-months in the prior one year.
* Self-reported diseases that could interfere with bone metabolism. For example, osteomalacia, bone cancer, myeloma, Pagets disease, hyper parathyroidism, hyperthyroidism not treated, severe renal (stage 4+ chronic kidney disease, history of dialysis, kidney transplant, etc.) or hepatic insufficiency, prolonged immobilization (more than 2 months in the previous year).
* If, in the opinion of a site PI, the subject is inappropriate for the scientific purposes of this study. For instance, a high fall risk patient due to an existing neurological disorder (e.g., Parkinsons disease, ALS, etc.) would be excluded.

Ages: 50 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: We will investigate and compare the abilities of OsteoDXs Cortical Bone Mechanics Technology (CBMT) and dual-energy x-ray absorptiometry (DXA) to discriminate between women ages 50-80 who have recently experienced a fragility fracture (n=138) and age-, BMI- and race-matched women who have not experienced a similar fracture (n=276 [1:2 allocation ratio]). Control subject matching will be done retrospectively with the goal being to match each case with controls that are within ~ 5 years, 3 BMI units, and of the same race.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Discriminatory Accuracy of CBMT vs. BMD | 1 Day
  Discriminatory accuracy of ulnar flexural rigidity in comparison to the bone mineral density.
CBMT's Added Value | 1 Day
  Binomial logistic regression's Walt coefficient to quantify how ulnar flexural rigidity and areal BMD predicts group membership (cases and controls).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Clark, PhD, Principal Investigator — Ohio Musculoskeletal and Neurological Institute (OMNI) at Ohio University
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Indiana Center for Musculoskeletal Health, Indianapolis, Indiana
  - Ohio Musculoskeletal and Neurological Institute at Ohio University, Athens, Ohio

IPD SHARING:
Plan to Share IPD: No